CLINICAL TRIAL: NCT02367105
Title: Testosterone Replacement to Augment Lifestyle Therapy in Obese Older Veterans
Brief Title: Lifestyle Intervention and Testosterone Replacement in Obese Seniors
Acronym: LITROS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Baylor College of Medicine (Other); Biomedical Research Institute of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ENDA-034-12F; CX000906 (Other Grant/Funding Number: VA CSRD)
Record Dates: First submitted 2015-01-21; First posted 2015-02-20 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-01

CONDITIONS: Obesity and Hypogonadism
Keywords: Obesity; Hypogonadism; Frailty
MeSH Terms: conditions — Obesity; Hypogonadism; Frailty | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone plus Lifestyle Therapy (Active Comparator): Testosterone replacement in combination with behavioral diet to induce ~10% weight loss + supervised aerobic and exercise training
  Interventions: Drug: Testosterone; Other: Lifestyle Therapy
- Placebo plus Lifestyle Therapy (Placebo Comparator): Placebo in combination with behavioral diet to induce ~10% weight loss and supervised aerobic and exercise training
  Interventions: Other: Lifestyle Therapy; Drug: Placebo

INTERVENTIONS:
Drug: Testosterone — Daily testosterone gel applied once daily in the morning to intact skin
  Arms: Testosterone plus Lifestyle Therapy
Other: Lifestyle Therapy — Weekly behavioral diet to induce ~10% weight loss in combination with supervised aerobic and exercise training three times a week
Drug: Placebo — Placebo gel for testosterone
  Arms: Placebo plus Lifestyle Therapy

SUMMARY:
The prevalence of obesity in Veterans is greater than in the general population, and even more so among users of the VA Health Care System. In addition, the population of obese older Veterans is rapidly increasing as more baby boomers become senior citizens. In older Veterans, obesity exacerbates the age- related decline in physical function and causes frailty which predisposes to admission to a VA chronic care facility. However, the optimal clinical approach to obesity in older adults is controversial because of the concern that weight loss therapy could be harmful by aggravating the age-related loss of muscle mass and bone mass. In fact, the MOVE (Managing Overweight/Obese Veterans) program does not have any guidelines for eligible Veterans if they are 70 or older. It is possible that the addition of testosterone replacement to lifestyle therapy will preserve muscle mass and bone mass and reverse frailty in obese older Veterans and thus prevent their loss of independence and decrease demand for VA health care services.

DETAILED DESCRIPTION:
Obesity is not only highly prevalent among Americans, but even more so among Veterans using VA medical facilities. Failure to assist Veterans in managing weight and sedentary lifestyle affects current treatment and increases future demand for VA health care services. Decreased muscle mass with aging and the need to carry extra mass due to obesity make it particularly difficult for obese older Veterans to function independently and results in frailty leading to increased nursing home admissions and increased morbidity and mortality. Data from preliminary studies showed that lifestyle therapy resulting in weight loss in this understudied population improves physical function and ameliorates frailty. However, this improvement in physical function is modest at best and most obese older adults remain physically frail. More importantly, there are concerns that lifestyle therapy may exacerbate underlying sarcopenia and osteopenia from weight loss- induced loss of lean body mass and bone mineral density (BMD). As a result, most geriatricians are reluctant to recommend lifestyle therapy that includes weight loss in obese frail elderly patients although the combination of weight loss and exercise is recommended as part of standard care for obese patients in general. Thus, it is not surprising that among Veterans, the MOVE (Managing Overweight/Obese Veterans) program does not have any guidelines for eligible Veterans if they are 70 or older. In addition to overeating and lack of exercise, age-related decline in anabolic hormone (i.e. testosterone) may contribute to sarcopenia and osteopenia, which in turn is exacerbated by obesity. Indeed, preliminary studies discovered that obese older men had markedly low levels of serum testosterone at baseline which remained low throughout the duration of lifestyle therapy. Because testosterone replacement therapy has been shown to increase muscle mass and BMD, it is therefore likely that concomitant testosterone replacement during lifestyle therapy in obese older adults would preserve lean body mass and BMD, and reverse frailty. Accordingly, the optimal management to the problem of sarcopenic obesity and frailty might require a comprehensive approach of a combination of lifestyle intervention and the correction of anabolic hormone deficiency. Therefore, the primary goal of this proposal is to conduct a randomized, comparative efficacy, double-blind, placebo-controlled (for testosterone) trial of the effects of 1) lifestyle therapy (1% diet-induced weight loss and exercise training) + testosterone replacement therapy versus 2) lifestyle therapy without testosterone replacement (testosterone placebo) in obese (BMI e 30 kg/m2) older (age e 65 yrs) male Veterans. The investigators hypothesize that 1) lifestyle therapy + testosterone replacement will cause a greater improvement in physical function than lifestyle therapy without concomitant testosterone replacement; 2) lifestyle therapy + testosterone replacement will cause a greater preservation of fat-free mass and thigh muscle volume than lifestyle therapy without testosterone replacement, 3) lifestyle therapy + testosterone replacement will cause a greater preservation in BMD and bone quality than lifestyle therapy without testosterone replacement, and 4) lifestyle therapy + testosterone replacement will cause a greater reduction in intramuscular proinflammatory cytokines than lifestyle therapy without testosterone replacement. The overarching hypothesis across aims is that a multifactorial intervention by means of lifestyle therapy plus testosterone replacement will be the most effective approach for reversing sarcopenic obesity and frailty in obese older male adults, as mediated by their additive effects in suppressing chronic inflammation, and stimulating muscle and bone anabolism. Obesity in older adults, including many aging Veterans, is a major public health problem. In fact, the public health success that has occurred in recent years could be in danger if lifestyles of older adults are neglected. The novel health outcomes and mechanistic-based data generated from this proposed randomized clinical trial (RCT) will have important ramifications for the standard of care for this rapidly increasing segment of the aging Veteran population.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be

* older (65-85 yr)
* obese (BMI 30 kg/m2 or greater) Veteran men with low testosterone (less than 300 mg/dL) as defined by the Endocrine Society
* mild to moderately frail
* must have stable weight (~not less than or more than 2 kg) during the last 6 months
* sedentary (regular exercise less than 1 h/week or less than 2x/week for the last 6 months)

Exclusion Criteria:

* Any major chronic diseases, or any condition that would interfere with exercise or dietary restriction, in which exercise or dietary restriction are contraindicated, or that would interfere with interpretation of results.
* Examples include, but are not limited to:

  * cardiopulmonary disease (e.g. recent myocardial infarction (MI), unstable angina, stroke etc) or unstable disease (e.g. CHF)
  * severe orthopedic/musculoskeletal or neuromuscular impairments
  * visual or hearing impairments
  * cognitive impairment (Mini Mental State Exam Score less than 24)
  * current use of bone active drugs
  * uncontrolled diabetes (i.e. fasting blood glucose more than 140 mg/dl and/or HbA1c greater than 9.5%).
* Any contraindications to testosterone supplementation

  * history of prostate or breast cancer
  * history of testicular disease
  * untreated sleep apnea
  * hematocrit more than 50%
  * prostate-related findings of palpable nodule on exam, a serum PSA of 4.0 ng/ml or greater
  * International Prostate Symptom Sore more than 19
  * history of venous thromboembolism
* Osteoporosis or a BMD T-score of -2.5 in the lumbar spine or total hip as well as those patients with a history of osteoporosis-related fracture (spine, hip, or wrist)

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Male
Enrollment: 83 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T Villareal, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Publications from this research will be made available to the public through the National Library of Medicine PubMed Central website within one year after the date of publication (guidance is provided on the ORD website).
  MEDVAMC will not provide unrestricted, open public access to large scale health related datasets because of re-identification concerns and the obligation to protect Veterans' private information. However, controlled public access will be provided to the greatest extent possible under specific DUAs or other written agreements, and open access will be provided to the final datasets underlying peer-reviewed publications (aggregated data that can be released with privacy and confidentiality risks).

REFERENCES:
- [Derived] Gregori G, Celli A, Barnouin Y, Paudyal A, Armamento-Villareal R, Napoli N, Qualls C, Villareal DT. Cognitive response to testosterone replacement added to intensive lifestyle intervention in older men with obesity and hypogonadism: prespecified secondary analyses of a randomized clinical trial. Am J Clin Nutr. 2021 Nov 8;114(5):1590-1599. doi: 10.1093/ajcn/nqab253. PMID 34375393

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through advertisements and review of medical records at the Michael E DeBakey VA Medical Center.
Pre-assignment Details: After obtaining written informed consent, potential participants underwent a comprehensive medical screening procedure, including an exercise stress test. If they were found eligible based on the inclusion/exclusion criteria, they were randomized into one of the two treatment groups.
Groups:
- Placebo + Lifestyle Therapy: Placebo in combination with behavioral diet to induce ~10% weight loss and supervised aerobic and exercise training
  Lifestyle Therapy: Weekly behavioral diet to induce ~10% weight loss in combination with supervised aerobic and exercise training three times a week
  Placebo: Placebo gel for testosterone
- Testosterone + Lifestyle Therapy: Testosterone replacement in combination with behavioral diet to induce ~10% weight loss + supervised aerobic and exercise training
  Testosterone: Daily testosterone gel applied once daily in the morning to intact skin
  Lifestyle Therapy: Weekly behavioral diet to induce ~10% weight loss in combination with supervised aerobic and exercise training three times a week
Period: Overall Study
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Started | 41 | 42
Completed | 36 | 34
Not Completed | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (3.2) | 73.6 (3.7) | 73.4 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 41 | 42 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was reported by the participants
  Participants
    Hispanic or Latino | 8 | 19 | 27
    Not Hispanic or Latino | 32 | 20 | 52
    Unknown or Not Reported | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was reported by the participants
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Black or African American | 14 | 20 | 34
    White | 22 | 19 | 41
    More than one race | 2 | 2 | 4
    Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 41 | 42 | 83
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — The body-mass index is the weight in kilograms divided by the square of the height in meters
  kg/m^2 | 36.9 (4.9) | 37.1 (5.6) | 37.0 (5.2)
Total testosterone level [Mean (Standard Deviation); unit: ng/dl] — Measured in the blood during early am in the fasting state.
  ng/dl | 218 (43) | 210 (63) | 214 (54)
Physical Performance Test score [Mean (Standard Deviation); unit: units on a scale] — The test includes walking 50 ft, putting on and removing a coat, picking up a penny, standing from a chair, lifting a book, climbing a flight of stairs, climbing up and down 4 flight of stairs, and performing a 360-degree turn. The score for each task ranges from 0 to 4; a perfect score is 36. Higher scores indicate better physical function.
  units on a scale | 28.3 (3.1) | 28.5 (2.8) | 28.4 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Physical Performance Test
Description: The primary functional outcome is the modified physical performance test, which includes seven standardized tasks (walking 50 ft, putting on and removing a coat, picking up a penny, standing up from a chair, lifting a book, climbing one flight of stairs, and performing a progressive Romberg tests) plus two additional tasks (climbing up and down four flights of stairs and performing a 360-degree turn). The score for each task ranges form 0 to 4; a perfect score is 36. Higher scores indicate better physical function.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
units on a scale | 4.6 (0.3) | 4.9 (0.3)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.58, Mixed Models Analysis; Baseline values as covariate; Mean Difference (Final Values) = -0.3

2. Secondary Outcome: Change in Endurance Capacity
Description: Assessed by measuring peak oxygen consumption using indirect calorimetry during a treadmill exercise stress test
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ml/kg/min
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
ml/kg/min | 2.8 (0.3) | 4.0 (0.3)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = 0.03, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = -1.2

3. Secondary Outcome: Change in Functional Status
Description: Assessed by the Functional Status Questionnaire. Score range: 0 to 36 with higher scores indicating better functional status
  Provides information of the participants ability to perform activities of daily living.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
units on a scale | 2.9 (0.4) | 3.1 (0.4)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = .97, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = 0.0

4. Secondary Outcome: Change in Body Weight
Description: Measured after an overnight fast using calibrated scales
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
kilograms | -10.6 (0.6) | -9.8 (0.6)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = 0.56, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = -0.7

5. Secondary Outcome: Change in Lean Body Mass
Description: Assessed by using dual-energy x-ray absorptiometry
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
kg | -2.4 (0.2) | -1.2 (0.2)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = 0.01, Mixed Models Analysis; Mean Difference (Final Values) = -1.2

6. Secondary Outcome: Change in Fat Mass
Description: Assessed by using dual-energy x-ray absorptiometry
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
kg | -8.2 (0.4) | -8.0 (0.5)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = 0.91, Mixed Models Analysis; Mean Difference (Final Values) = -1.1

7. Secondary Outcome: Change in Thigh Muscle Volume
Description: Assessed by using magnetic resonance imaging
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: cm^3
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
cm^3 | -68 (10) | -25 (10)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy; Test type: Superiority; p = 0.04, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = -42

8. Secondary Outcome: Thigh Fat Volume
Description: Volume of fat in the thigh by measured by magnetic resonance imaging
Time Frame: 6 months
Measure: Mean (Standard Error); unit: cm^3
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
cm^3 | -292 (31) | -262 (32)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = .67, Mixed Models Analysis; Baseline values as covariates; Mean Difference (Final Values) = -29

9. Secondary Outcome: Change in Total Hip Bone Mineral Density
Description: Assessed by using dual-energy x-ray absorptiometry
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: gm/cm^2
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
gm/cm^2 | -0.013 (0.002) | 0.007 (0.002)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = 0.003, Mixed Models Analysis; Baseline valued adjusted; Mean Difference (Final Values) = -0.019

10. Secondary Outcome: Change in Lumbar Spine Bone Mineral Density
Description: As measured by Dual energy x-ray absorptiometry
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: gm/cm^2
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
gm/cm^2 | 0.004 (0.004) | 0.007 (0.004)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = 0.69, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = -0.003

11. Secondary Outcome: Change in Muscle Strength
Description: assessed by total1-repetition maximum (the maximal weight lifted at one time; the totals are the sum of the maximal weights lifted in the biceps curl, bench press, 387 seated row, knee extension, knee flexion, and leg press exercises).
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
kg | 72 (5) | 68 (5)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = 0.94, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = 7

12. Secondary Outcome: Change in Static Balance
Description: assessed by one leg limb stance
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
seconds | 4.5 (0.9) | 5.0 (0.9)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.41, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = -0.5

13. Secondary Outcome: Change in Dynamic Balance
Description: Assessed by using the obstacle course
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Testosterone Plus Lifestyle Therapy | Placebo Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
seconds | -2.9 (0.3) | -3.2 (0.4)
Statistical Analysis 1: Comparison: Testosterone Plus Lifestyle Therapy vs Placebo Plus Lifestyle Therapy; Test type: Superiority; p = 0.46, Mixed Models Analysis; Baseline values as covariates; Mean Difference (Final Values) = 0.5

14. Secondary Outcome: Change in Gait Speed
Description: Determined by measuring the time needed to walk 25 ft.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: m/min
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
m/min | 8.6 (1.3) | 8.2 (1.4)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority — Baseline value adjusted; p = 0.96, Mixed Models Analysis; Mean Difference (Final Values) = 0.6

15. Secondary Outcome: Change in Composite Cognitive Z-score
Description: Test of overall cognitive performance formed by averaging the standardized scores for several domains of cognitive function (attention, memory, executive, language, global). Higher scores indicate better cognitive status.
  The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of the baseline scores (units on a scale). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
z-score | .273 (.061) | .557 (.065)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = .003, Mixed Models Analysis; Mean Difference (Final Values) = -.284

16. Secondary Outcome: Change in Modified Mini-mental Exam
Description: Test of global cognition with components for orientation, registration, attention, language, praxis, and immediate and delayed memory. Score ranges from 0 to 100 with higher scores indicate better cognition.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
units on a scale | 1.2 (0.3) | 2.1 (0.3)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = .16, Mixed Models Analysis; Baseline value and years of education as covariates; Mean Difference (Final Values) = -0.9

17. Secondary Outcome: Stroop Interference
Description: Assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect.
  Minimum score is 0, there is no maximum value. Higher scores indicate better outcome.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
score on a scale | 4.6 (0.7) | 3.1 (0.7)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = 0.21, Mixed Models Analysis; Baseline values and years of education as covariates; Mean Difference (Final Values) = -1.8

18. Secondary Outcome: Change in Word List Fluency
Description: Measure of verbal production, semantic memory, and language. Minimum score is 0, there is no maximum value. Higher scores indicate better outcome.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
units on a scale | 0.2 (0.5) | 0.9 (0.5)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = 0.41, Mixed Models Analysis; Baseline values and years of education as covariates; Mean Difference (Final Values) = -0.8

19. Secondary Outcome: Change in Ray Auditory Verbal Learning Test
Description: The Rey Auditory Verbal Learning Test (RAVLT) evaluates a wide diversity of functions: short-term auditory-verbal memory, rate of learning, learning strategies, retroactive, and proactive interference, presence of confabulation of confusion in memory processes, retention of information.
  Minimum score is 0, there is no maximum value. Higher scores indicate better outcome.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
units on a scale | 3.1 (0.9) | 7.0 (1.0)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = .03, Mixed Models Analysis; Baseline value and years if education as covariates; Mean Difference (Final Values) = -4.0

20. Secondary Outcome: Change in Trail A
Description: Test of visuospatial scanning, speed of processing, mental flexibility, and executive function (with a greater focus on attention).
  Minimum score is 0, there is no maximum value. Higher scores indicate better outcome.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
units on a scale | -7.7 (1.4) | -13.9 (1.5)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = .03, Mixed Models Analysis; Baseline values and years of education as covariates; Mean Difference (Final Values) = 6.6

21. Secondary Outcome: Change in Trail B
Description: Test of visuospatial scanning, speed of processing, mental flexibility, and executive function (with a focus on executive function)
  Minimum score is 0, there is no maximum value. Higher scores indicate better outcome.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
units on a scale | -10.2 (2.9) | -19.5 (3.0)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = .18, Mixed Models Analysis; Baseline values and years of education as covariates; Mean Difference (Final Values) = 7.8

22. Secondary Outcome: Change in Symbol Digital Modalities Test
Description: Assesses key neurocognitive functions that underlie many substitution tasks, including attention, visual scanning, and motor speed.
  Minimum score is 0, there is no maximum value. Higher scores indicate better outcome.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
units on a scale | 1.1 (0.5) | 2.8 (0.5)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.10, Mixed Models Analysis; Baseline values and years of education as covariates; Mean Difference (Final Values) = -1.7

23. Secondary Outcome: Change in Trabecular Bone Score
Description: The trabecular bone score is a measure of bone texture correlated with bone microarchitecture and a marker for the risk of osteoporosis.
  Minimum score is 0, there is no maximum value. Higher scores indicate better bone microarchitecture.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
units on a scale | 0.12 (.01) | .11 (.01)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = .65, Mixed Models Analysis; Baseline values as covariates; Mean Difference (Final Values) = .01

24. Secondary Outcome: Change in C-terminal Telopeptide
Description: biochemical marker of bone turnover (bone resorption) as measured by immunoassay technique
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: µg/L
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
µg/L | 0.530 (.012) | 0.002 (0.012)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy; Test type: Superiority; p = 0.03, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = 0.553

25. Secondary Outcome: Change in N-terminal Propeptide of Type I Procollagen
Description: Biochemical marker of bone turnover (bone formation) as measured by radioimmunoassay technique
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: µg/L
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
µg/L | -4.7 (1.4) | 1.5 (1.5)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.04, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = -6.5

26. Secondary Outcome: Change in Insulin Growth Factor-1
Description: Measured by immunoassay methodology
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
ng/mL | 11.8 (2.8) | 16.9 (3.0)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.35, Mixed Models Analysis — Baseline value adjusted; Mean Difference (Final Values) = 5.5

27. Secondary Outcome: Change in Trabecular Bone Score (Trabecular Bone Quality)
Description: assessed by trabecular bone score (TBS), a newly developed index for assessing trabecular bone quality and fracture risk.
  TBS is a bone texture parameter that quantifies cancellous bone microachitecture, which is key in determining bone strength and resistance to fracture, by computing raw data from dual energy x-ray absorptiometry of the lumbar spine.
  There are no minimum or maximum values. Higher scores mean better outcome.
Time Frame: Baseline and 6 months
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Testosterone + Lifestyle Therapy | Placebo + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
units on a scale | 0.11 (.01) | 0.12 (.01)
Statistical Analysis 1: Comparison: Testosterone + Lifestyle Therapy vs Placebo + Lifestyle Therapy; Test type: Superiority; p = 0.65, Mixed Models Analysis; Baseline value adjusted; Median Difference (Final Values) = 0.01

28. Secondary Outcome: Change in Levels of 25-hydroxyvitamin D
Description: assessed by using immunoassay methodology
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
ng/mL | 6.2 (1.1) | 8.3 (1.2)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.27, Mixed Models Analysis — Baseline value adjusted; Mean Difference (Final Values) = -2.4

29. Secondary Outcome: Change in Parathyroid Hormone Level
Description: Measured by immunoassay methodology as marker of bone metabolism
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
pg/mL | 12.9 (2.0) | 9.0 (2.0)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.39, Mixed Models Analysis — Baseline value adjusted; Mean Difference (Final Values) = -3.6

30. Secondary Outcome: Change in High-sensitivity C-reactive Protein (Inflammatory Marker)
Description: measured in the peripheral blood using immunoassay technique methodology
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
mg/dl | .19 (.05) | .18 (.05)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.58, Mixed Models Analysis; Mean Difference (Final Values) = .01

31. Secondary Outcome: Change in Interleukin-6
Description: Measured from fasting serum using immunoassay technique as marker of inflammation
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
pg/mL | -1.1 (0.2) | -1.0 (0.2)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.90, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = 0.1

32. Other Pre Specified Outcome: Change in Total Testosterone Levels
Description: as measured in the peripheral blood by liquid chromatography/mass spectrometry
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
ng/dL | 60 (21) | 306 (23)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = -252

33. Other Pre Specified Outcome: Change in Estradiol
Description: As measured by LC-MS/MS
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: pg/dL
Arm/Group | Testosterone + Lifestyle Therapy | Placebo + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
pg/dL | -3.0 (2.7) | 22.1 (2.9)
Statistical Analysis 1: Comparison: Testosterone + Lifestyle Therapy vs Placebo + Lifestyle Therapy; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline value as covariates; Mean Difference (Final Values) = -24.9

34. Other Pre Specified Outcome: Change in Hematocrit
Description: the ratio of the volume of red blood cells to the total volume of blood.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: percentage of red blood cells
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
percentage of red blood cells | -0.5 (0.3) | 2.4 (0.4)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p < 0.001, Mixed Models Analysis; Baseline values as covariates; Mean Difference (Final Values) = -2.7

35. Other Pre Specified Outcome: Change in Prostate Specific Antigen
Description: blood test to screen for prostate cancer
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
ng/mL | 0.2 (0.1) | 0.5 (0.1)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = 0.31, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = -0.2

36. Other Pre Specified Outcome: Change in Short Form Health Survey (SF-36) Quality of Life Physical Component
Description: Using Short Form-36 of Life Questionnaire Physical Component subscale. Minimum score is 0, Maximum score is 100. Higher scores indicate better outcome.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
units on a scale | 5.5 (0.8) | 7.1 (0.8)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = 0.42, Mixed Models Analysis — Baseline values as covariates; Mean Difference (Final Values) = -1.2

37. Other Pre Specified Outcome: Change in International Prostate Symptom Score
Description: Using the International Prostate Symptom Scoring (IPS); Minimum score is 0, Maximum score is 35. Higher scores mean worse outcome.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
units on a scale | -0.2 (0.5) | -0.1 (0.5)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.69, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = -0.4

38. Other Pre Specified Outcome: Change in Triglyceride Levels
Description: Blood samples obtained in the fasting state as part of measurements of lipid profile
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
mg/dl | -39 (5.4) | -31 (5.0)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.23, Mixed Models Analysis; Baseline value adjusted; Mean Difference (Final Values) = -13.1

39. Other Pre Specified Outcome: Change in HDL-cholesterol
Description: Blood samples obtained in the fasting state as part of measurements of lipid profile
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
mg/dl | 5.4 (1.0) | 0.2 (1.1)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.01, Mixed Models Analysis; Mean Difference (Final Values) = 5.3

40. Other Pre Specified Outcome: Change in Waist Circumference
Description: Waist circumference as measured horizontally at the midpoint between the highest point of the iliac crest and the lowest portion of the 12th rib in the standing position.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: cm
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
cm | -9.4 (0.5) | -8.4 (0.6)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = 0.36, Mixed Models Analysis; Baseline values as covariates; Mean Difference (Net) = -1.0

41. Other Pre Specified Outcome: Change in Glucose
Description: Measured in the blood after overnight fast
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
mg/dl | -22.5 (3.7) | -17.1 (3.8)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy vs Testosterone Plus Lifestyle Therapy; Test type: Superiority; p = 0.23, Mixed Models Analysis; Baseline values as covariates; Mean Difference (Final Values) = -8.6

42. Other Pre Specified Outcome: Change in Mood
Description: Using Yesavage Depression Scale Lower scores indicate better mood (range 0 to 30).
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
score on a scale | -1.43 (0.38) | -1.39 (0.39)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.69, Mixed Models Analysis; Baseline values adjusted; Mean Difference (Final Values) = -0.31

43. Other Pre Specified Outcome: Number of Participants With Significant Changes in Functional Connectivity in the Default Mode Network
Description: Functional connectivity was measured with seeds of the DMN (medial prefrontal cortex [MPFC] and posterior cingulate cortex [PCC]). Correlation coefficients representing the degree of connectivity between hypothesized regions were Fisher transformed. An a priori threshold of p<.001 at the voxel level and p<.05, FDR corrected for multiple comparisons across the whole brain, at the cluster level were used to determine significant connectivity.
Time Frame: Baseline and 6 months
Population: The number of subjects per group is less than the overall number of subjects enrolled in the trial because this was an add-on outcome later in the study. Moreover, the analyses are limited to subjects with complete evaluable pre and post-MRI data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 6 | 11
Participants
  DMN (MPFC seed) | 0 | 0
  DMN (PCC seed) | 0 | 0
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy vs Testosterone + Lifestyle Therapy; Test type: Superiority; p > .05, t-test, 2 sided — A priori threshold = voxel p<.001, cluster p<.05, false discovery rate (FDR) whole brain correction. There is no correction for multiple seeds given small sample sizes and pre-post design; Number of participants = 0

44. Other Pre Specified Outcome: Change in Skeletal Muscle Growth Factor (MYOD1)
Description: Assessed by using RNA-seq quantification of gene expression in skeletal muscles obtained during muscle biopsies.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: log2fold
Arm/Group | Placebo Plus Lifestyle Therapy | Testosterone Plus Lifestyle Therapy
Number analyzed (Participants) | 20 | 18
log2fold | 0.23 (0.05) | 0.53 (0.12)
Statistical Analysis 1: Comparison: Placebo Plus Lifestyle Therapy; 6 months vs Baseline; Test type: Superiority; p = 0.37, t-test, 2 sided — Using DESeq2 R package. P values were adjusted using the Benjamini and Hochberg's approach for controlling the false discovery rate; Mean Difference (Net) = 0.23, Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Testosterone Plus Lifestyle Therapy; 6 months vs Baseline; Test type: Superiority; p = .02, t-test, 2 sided — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = 0.58, Standard Error of Mean 0.12

45. Other Pre Specified Outcome: Change in Peripheral Quantitative Computed Tomography Measures (Volumetric Bone Density)
Description: assessed by quantitative computed tomography at 4% distal tibia using the following thresholds: 180 mg/cm3 and 45% of the area
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mg/cm^3
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
Number analyzed (Participants) | 41 | 42
mg/cm^3 | -3.1 (1.3) | -0.3 (1.3)
Statistical Analysis 1: Comparison: Placebo + Lifestyle Therapy; Test type: Superiority; p = .05, Mixed Models Analysis; Final vs baseline; Mean Difference (Net) = -0.3, Standard Error of Mean 1.3
Statistical Analysis 2: Comparison: Testosterone + Lifestyle Therapy; Test type: Superiority; p = 0.3, Mixed Models Analysis; Final vs baseline; Mean Difference (Net) = -0.3, Standard Error of Mean 1.3

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo + Lifestyle Therapy | Testosterone + Lifestyle Therapy
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/42
Other Adverse Events (participants affected / at risk) | 12/41 | 6/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Lifestyle Therapy (N=41) | Testosterone + Lifestyle Therapy (N=42)
Congestive heart failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bleeding peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Idiopathic thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyperosmolar hyperglycemic state (Endocrine disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Lifestyle Therapy (N=41) | Testosterone + Lifestyle Therapy (N=42)
hypoglycemia, asymptomatic and symptomatic (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Elevated PSA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Dizziness/orthostasis (Vascular disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/05/NCT02367105/Prot_SAP_000.pdf